CLINICAL TRIAL: NCT07383376
Title: Investigation of the Functional, Aesthetic, and Quality-of-life Effects of Combined Surgical-orthodontic Treatment
Brief Title: Investigation of Skeletally Anchored Expansion of the Maxilla
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SE RKEB 249/2024
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Palatal Expansion Technique
Keywords: maxillary expansion; orthodontics; occlusion
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Intervention Model Description: PICO
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgically Assisted Rapid Maxillary Expansion (Active Comparator): Participants in this arm will undergo surgically assisted rapid palatal expansion (SARPE). The procedure will include surgical weakening of the maxillary sutures followed by maxillary expansion using a palatal expansion appliance. The appliance will be activated according to a standardized protocol. Clinical and radiographic assessments will be performed to evaluate treatment outcomes.
  Interventions: Procedure: SARME
- Non-Surgically Assisted Rapid Maxillary Expansion (Experimental): Participants in this arm will undergo non-surgical maxillary expansion using a miniscrew-assisted rapid palatal expansion (MARPE) appliance. The appliance will be anchored to the palate using temporary anchorage devices (TADs) and activated according to a standardized expansion protocol. No surgical assistance will be performed in this group. Clinical and radiographic assessments will be used to evaluate treatment outcomes.
  Interventions: Device: MARPE

INTERVENTIONS:
Device: MARPE — Miniscrew-assisted rapid palatal expander (MARPE)
  Arms: Non-Surgically Assisted Rapid Maxillary Expansion
Procedure: SARME — Surgically assisted rapid palatal expansion (SARPE).
  Arms: Surgically Assisted Rapid Maxillary Expansion

SUMMARY:
This study aims to compare two different methods for maxillary expansion in adult patients with transverse maxillary deficiency. Participants will receive either miniscrew-assisted rapid palatal expansion (MARPE-MICRO-4). We want to compare the surgically assisted rapid palatal expansion (SARPE) and the non surgical/conservative method. Clinical (3D scans of the upper jaws) measurements will be used to evaluate skeletal expansion and stability over time. Approximately 40 adult patients will be included and followed for 12 months. The results of this study may help clinicians choose the most appropriate treatment method for adult maxillary expansion.

ELIGIBILITY:
Inclusion Criteria:

* Presence of transverse maxillary deficiency requiring maxillary expansion
* Indication for either non-surgical (MARPE) or surgically assisted (SARPE) maxillary expansion
* Permanent dentition
* Ability to understand the study procedures and provide informed consent

Exclusion Criteria:

* Previous maxillary expansion treatment
* Craniofacial syndromes or cleft lip/palate
* Severe periodontal disease
* Active oral infection
* Systemic conditions affecting bone metabolism
* Pregnancy or breastfeeding
* Inability to comply with study procedures or follow-up visits

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Skeletal maxillary expansion measured with 3D scans | Baseline to 6 months after completion of maxillary expansion.
  Changes in intermolar and intercanine width will be measured on digital dental models.

SECONDARY OUTCOMES:
Buccal tipping of posterior teeth measured on 3D digital models | Baseline to 6 months after completion of maxillary expansion
  Buccal tipping of posterior teeth will be assessed using 3D digital dental models by measuring changes in crown inclination of maxillary premolars and molars before treatment and after completion of maxillary expansion.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatric Dentistry and Orthodontics, Semmelweis University, Budapest, Pest County, Hungary

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared upon reasonable request after publication of the primary results. Requests will be reviewed by the study investigators and data will be provided in accordance with institutional and ethical regulations.
Supporting Information: Study Protocol
Time Frame: De-identified individual participant data and the study protocol will be available after publication of the primary results and will remain available for 5 years.
Access Criteria: Access to de-identified individual participant data and supporting documents will be provided to qualified researchers upon reasonable request. Requests will be reviewed by the study investigators and data will be shared in accordance with institutional policies and ethical approvals.